CLINICAL TRIAL: NCT02555358
Title: Three Drugs in Advanced Gastric Cancer Neoadjuvant Chemotherapy for Stage Ⅲ Multicenter, Open, Randomized, Controlled Clinical Study
Brief Title: Three Drugs in Advanced Gastric Cancer Neoadjuvant Chemotherapy for Stage Ⅲ Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qun Zhao (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Qun Zhao, Surgical director, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Alien Craft 0004
Record Dates: First submitted 2015-07-22; First posted 2015-09-21 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
Keywords: Resectable advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A（DOX） (Experimental): Interventions：This arm wil receive four cycles of DOX (docetaxel 60mg/m2 on day 1,oxaliplatin 130mg/m2 on day 1 and capecitabine 1,000 mg/m2 per day on days 1 to 14, repeated every 3 weeks) as neoadjuvant therapy and four cycles of Xelox (capecitabine 1,000 mg/m2 per day on days 1 to 14 and oxaliplatin 130mg/m2 on day 1, repeated every 3 weeks) as adjuvant therapy
  Interventions: Drug: docetaxel,0xaliplatin,capecitabine
- B（Xelox） (Active Comparator): Interventions：This arm wil receive four cycles of Xelox (capecitabine 1,000 mg/m2 per day on days 1 to 14 and oxaliplatin 130mg/m2 on day 1, repeated every 3 weeks) as neoadjuvant therapy and four cycles of Xelox as adjuvant therapy
  Interventions: Drug: oxaliplatin,capecitabine
- C（Xelox） (Active Comparator): Interventions：This arm wil receive eight cycles of Xelox (capecitabine 1,000 mg/m2 per day on days 1 to 14 and oxaliplatin 130mg/m2 on day 1, repeated every 3 weeks) as adjuvant therapy.
  Interventions: Drug: oxaliplatin,capecitabine

INTERVENTIONS:
Drug: docetaxel,0xaliplatin,capecitabine — docetaxel 60mg/m2， ivgtt，2h，d1;capecitabine 1000mg/m2 po bid d1-14; oxaliplatin 130mg/m2， ivgtt，2h，d1;q21d
  Other Names: AISU,AIHENG,AIBIN
  Arms: A（DOX）
Drug: oxaliplatin,capecitabine — oxaliplatin 130mg/m2， ivgtt，2h，d1;capecitabine 1000mg/m2 po bid d1-14;q21d
  Other Names: AIHENG,AIBIN
  Arms: B（Xelox）; C（Xelox）

SUMMARY:
The purpose of this study is to assess the relationship of pCR rate and efficacy by comparing the two drugs and three drugs as neoadjuvant chemotherapy in advanced gastric cancer patients.

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned by a randomisation system in a 1:1:1 ratio to three group. The group A wil receive four cycles of DOX (docetaxel 60mg/m2 on day 1,oxaliplatin 130mg/m2 on day 1 and capecitabine 1,000 mg/m2 per day on days 1 to 14, repeated every 3 weeks) as neoadjuvant therapy and four cycles of Xelox (capecitabine 1,000 mg/m2 per day on days 1 to 14 and oxaliplatin 130mg/m2 on day 1, repeated every 3 weeks) as adjuvant therapy.The group B wil receive four cycles of Xelox (capecitabine 1,000 mg/m2 per day on days 1 to 14 and oxaliplatin 130mg/m2 on day 1, repeated every 3 weeks) as neoadjuvant therapy and four cycles of Xelox as adjuvant therapy.The group C wil receive eight cycles of Xelox (capecitabine 1,000 mg/m2 per day on days 1 to 14 and oxaliplatin 130mg/m2 on day 1, repeated every 3 weeks) as adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven in operable advanced gastric adenocarcinoma;
2. Subjects who were identified as potentially resectable cases by a multidisciplinary consultation;
3. KPS> 80; ECOG score: 0-1;
4. Expected survival> 6 months;
5. Age 20 -60;
6. Major organ function has to meet the following criteria:

   Neutrophil count ≥1.5 × 109 / L, platelet count ≥100 × 109 / L, Hemoglobin ≥90g / L, liver function <1.5 times the upper limit of normal, serum bilirubin ≤1.0 × UNL, serum creatinine <1.5 × UNL, PT-INR / PTT <1.7 times the upper limit of normal;
7. Subjects has to voluntarily join the study and sign the Informed Consent Form for the study;

Exclusion Criteria:

1. Associated with serious diseases in liver ,kidney, cardiovascular system and other vital organs;
2. History of hypersensitivity to docetaxel, capecitabine, oxaliplatin or the ingredients of this product;
3. Receiving any form of chemotherapy or other study medication;
4. Pregnancy or lactation women, or women with suspected pregnancy or men unless using a reliable and appropriate contraceptive method;
5. Associated with inability to swallow, haemorrhagic peptic ulcer, mechanical or paralytic ileus, gastrointestinal active bleeding.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-11; Primary Completion 2021-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
The pathological complete response rate | 24 weeks

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
Progression-free survival(PFS) | 3 years
Disease-free survival(DFS) | 3 years
Adverse events | 3 years
  Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, version 2.0. The number of Participants with adverse events will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, director, Study Chair — The 4th Hospital of Hebei Medical University
Locations (1):
- Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Result] 1. Zhao Q, Li Y, Tan BB, Tian Y, Jiao ZK, Zhao XF, Zhang ZD, Wang D, Yang PG. XELOX neoadjuvant chemotherapy for advanced gastric cancer resection rate and the impact on prognosis. Journal of Cancer 2013,35 (10) : 773-777 2. Zhao Q, Li Y, Wang GY, Jiao ZK, Zhao XF, Zhang ZD, Tan BB, Zhou CX, Sun WL laparoscopic abdominal control study of gastric cancer resection surgery clinical effect. Chinese General Practice, 2013,16 (1B): 210-215. 3.Zhao Q, Li Y, Tian Y, Chen YN, Tan BB, Zhao XF, Jiao ZK, Zhang ZD, Chang SL. Histological Complete Response after Neoadjuvant XELOX in Advanced Gastric Carcinoma. Hepatogastroenterology. 2013 Jan 24;60(126)
- [Derived] Tian Y, Yang P, Guo H, Liu Y, Zhang Z, Ding P, Zheng T, Deng H, Ma W, Li Y, Fan L, Zhang Z, Wang D, Zhao X, Tan B, Liu Y, Zhao Q. Neoadjuvant docetaxel, oxaliplatin plus capecitabine versus oxaliplatin plus capecitabine for patients with locally advanced gastric adenocarcinoma: long-term results of a phase III randomized controlled trial. Int J Surg. 2023 Dec 1;109(12):4000-4008. doi: 10.1097/JS9.0000000000000692. PMID 37678277